CLINICAL TRIAL: NCT05585307
Title: An Umbrella Phase 1b, Open-label, Multi-Cohort Study to Evaluate Safety, Pharmacokinetics, and Antiviral Activity of Novel Antiretrovirals in Participants With HIV-1
Brief Title: Study of Novel Antiretrovirals in Participants With HIV-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-544-5905
Record Dates: First submitted 2022-10-14; First posted 2022-10-18 (Actual); Results first posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination; Standard of Care

STUDY DESIGN:
Intervention Model Description: The Substudies were conducted in parallel. However, the cohorts within the Substudies received drug assignment sequentially.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Substudy 01: Cohort 1: Bavtavirine 675 mg (High-Fat Meal) (Experimental): Participants receive a single dose of bavtavirine 675 mg tablet with a high-fat meal on Day 1. After assessments on Day 11 or upon early termination (ET), the participants initiate a regimen of B/F/TAF, or an alternative standard of care (SOC) antiretroviral (ART) regimen (example INSTI + NRTIs: dolutegravir (DTG)/abacavir (ABC)/3TC or DTG/3TC) up to Day 39.
  Interventions: Drug: Bavtavirine; Drug: B/F/TAF; Drug: Standard of Care (Substudy 01)
- Substudy 01: Cohort 2: Bavtavirine 1200 mg (Low-Fat Meal) (Experimental): Participants receive a single dose of bavtavirine 1200 mg tablet with a low-fat meal on Day 1. After assessments on Day 11 or upon ET, the participants initiate a regimen of B/F/TAF, or an alternative SOC ART regimen (example INSTI + NRTIs: DTG/ABC/3TC or DTG/3TC) up to Day 39.
  Interventions: Drug: Bavtavirine; Drug: B/F/TAF; Drug: Standard of Care (Substudy 01)
- Substudy 01: Cohort 3: Bavtavirine 900 mg (High-Fat Meal) (Experimental): Participants receive bavtavirine 900 mg tablet with a high-fat meal on Days 1 and 2. After assessments on Day 11 or upon ET, the participants initiate a regimen of B/F/TAF, or an alternative SOC ART regimen (example INSTI + NRTIs: DTG/ABC/3TC or DTG/3TC) up to Day 39.
  Interventions: Drug: Bavtavirine; Drug: B/F/TAF; Drug: Standard of Care (Substudy 01)
- Substudy 02: Cohort 1: GS-1720 450 mg (Experimental): Participants receive a single dose of GS-1720 450 mg tablet on both Days 1 and 2 in fasted condition. After assessments on Day 11 or upon ET, the participants initiate a regimen of B/F/TAF, or an alternative SOC ART regimen (example INSTI + NRTIs: DTG/ABC/3TC or DTG/3TC) up to Day 60.
  Interventions: Drug: B/F/TAF; Drug: GS-1720; Drug: Standard of Care (Substudy 02)
- Substudy 02: Cohort 2: GS-1720 150 mg (Experimental): Participants receive a single dose of GS-1720 150 mg tablet on both Days 1 and 2 in fasted condition. After assessments on Day 11 or upon ET, the participants initiate a regimen of B/F/TAF, or an alternative SOC ART regimen (example INSTI + NRTIs: DTG/ABC/3TC or DTG/3TC) up to Day 60.
  Interventions: Drug: B/F/TAF; Drug: GS-1720; Drug: Standard of Care (Substudy 02)
- Substudy 02: Cohort 3: GS-1720 30 mg (Experimental): Participants receive a single dose of GS-1720 30 mg tablet on both Days 1 and 2 in fasted condition. After assessments on Day 11 or upon ET, the participants initiate a regimen of B/F/TAF, or an alternative SOC ART regimen (example INSTI + NRTIs: DTG/ABC/3TC or DTG/3TC) up to Day 60.
  Interventions: Drug: B/F/TAF; Drug: GS-1720; Drug: Standard of Care (Substudy 02)
- Substudy 02: Cohort 4: GS-1720 900 mg (Experimental): Participants receive a single dose of GS-1720 900 mg tablet on both Days 1 and 2 in fasted condition. After assessments on Day 11 or upon ET, the participants initiate a regimen of B/F/TAF, or an alternative SOC ART regimen (example INSTI + NRTIs: DTG/ABC/3TC or DTG/3TC) up to Day 60.
  Interventions: Drug: B/F/TAF; Drug: GS-1720; Drug: Standard of Care (Substudy 02)
- Substudy 03: Cohort 1: GS- 6212 100 mg (Experimental): Participants receive GS-6212 100 mg tablet twice daily on Days 1 through 10. After assessments on Day 11 or upon ET, the participants initiate a regimen of B/F/TAF, or an alternative SOC ART regimen (example INSTI + NRTIs: DTG/ABC/3TC or DTG/3TC) up to Day 25.
  Interventions: Drug: B/F/TAF; Drug: GS-6212; Drug: Standard of Care (Substudy 03)

INTERVENTIONS:
Drug: Bavtavirine — Administered orally
  Other Names: GS-5894
  Arms: Substudy 01: Cohort 1: Bavtavirine 675 mg (High-Fat Meal); Substudy 01: Cohort 2: Bavtavirine 1200 mg (Low-Fat Meal); Substudy 01: Cohort 3: Bavtavirine 900 mg (High-Fat Meal)
Drug: B/F/TAF — Administered orally
  Other Names: Biktarvy®
Drug: Standard of Care (Substudy 01) — Antiretroviral therapy, administered orally
  Non-NNRTIs, examples: ABC/DTG/3TC; DTG plus (TAF or TDF) plus (FTC or 3TC)
  Arms: Substudy 01: Cohort 1: Bavtavirine 675 mg (High-Fat Meal); Substudy 01: Cohort 2: Bavtavirine 1200 mg (Low-Fat Meal); Substudy 01: Cohort 3: Bavtavirine 900 mg (High-Fat Meal)
Drug: GS-1720 — Administered orally
  Arms: Substudy 02: Cohort 1: GS-1720 450 mg; Substudy 02: Cohort 2: GS-1720 150 mg; Substudy 02: Cohort 3: GS-1720 30 mg; Substudy 02: Cohort 4: GS-1720 900 mg
Drug: Standard of Care (Substudy 02) — Antiretroviral therapy, administered orally
  Example INSTIs: DTG/ABC/3TC or DTG/3TC
  Arms: Substudy 02: Cohort 1: GS-1720 450 mg; Substudy 02: Cohort 2: GS-1720 150 mg; Substudy 02: Cohort 3: GS-1720 30 mg; Substudy 02: Cohort 4: GS-1720 900 mg
Drug: GS-6212 — Administered orally
  Arms: Substudy 03: Cohort 1: GS- 6212 100 mg
Drug: Standard of Care (Substudy 03) — Antiretroviral therapy, administered orally
  Arms: Substudy 03: Cohort 1: GS- 6212 100 mg

SUMMARY:
Master protocol: The goal of this master clinical trial study is to learn how novel antiretrovirals (medicines that stop the virus from multiplying) affect the human immunodeficiency virus-1 (HIV-1) infection in people living with HIV (PWH).

Substudy-01 (GS-US-544-5905-01) will evaluate bavtavirine in PWH.

Substudy-02 (GS-US-544-5905-02) will evaluate GS-1720 in PWH.

Substudy-03 (GS-US-544-5905-03) will evaluate GS-6212 in PWH.

DETAILED DESCRIPTION:
This umbrella study will begin with a substudy of bavtavirine (Substudy-01), and later substudies GS-1720 (Substudy-02) and GS-6212 (Substudy-03) will be added. Substudies evaluating additional study drugs will be added in a staggered manner when relevant nonclinical and/or clinical data become available.

* Substudy-01 enrollment closed, actual enrollment is 13.
* Substudy-02 enrollment closed, actual enrollment is 28.
* Substudy-03 enrollment closed, actual enrollment is 8.

ELIGIBILITY:
Key Inclusion Criteria:

All Substudies:

* Plasma human immunodeficiency virus-1 (HIV-1) ribonucleic acid (RNA) ≥ 5000 copies/mL but ≤ 400,000 copies/mL at screening.
* Cluster of differentiation 4 (CD4) cell count > 200 cells/mm^3 at screening.
* Antiretroviral (ARV) treatment-naive or treatment-experienced but naive to the investigational ARV drug class being investigated in the given substudy and have not received any ARV within 12 weeks of screening, including medications received for pre-exposure prophylaxis (PrEP) or postexposure prophylaxis (PEP) (note that current or prior receipt of long acting (LA) parenteral ARVs such as monoclonal antibodies (mAbs) targeting HIV-1, injectable cabotegravir (CAB), or injectable rilpivirine (RPV) is exclusionary).
* Have adequate renal function (estimated glomerular filtration rate (eGFR) ≥ 70 mL/min/1.73 m^2)
* No clinically significant abnormalities in electrocardiogram (ECG) at screening.

Substudy-01, Substudy-02, and Substudy-03:

* Participants in substudy-01 should be willing to initiate a non-NNRTI based SOC ART on Day 11.
* Participants in substudy-02 and Substudy-03 should be willing to initiate any SOC ART on Day 11.
* Willing and able to comply with meal requirements on dosing days.

Key Exclusion Criteria:

All Substudies:

* Known historical genotypic or phenotypic resistance to 4 major ARV classes (nucleoside reverse transcriptase inhibitor (NRTI), nonnucleoside reverse transcriptase inhibitor (NNRTI), protease inhibitor (PI), integrase strand-transfer inhibitor (INSTI)).
* History of an AIDS-defining condition including present at the time of screening.
* Active, serious infections (other than HIV-1) requiring therapy and including active tuberculosis infection < 30 days prior to randomization.
* History of or current clinical decompensated liver cirrhosis (eg, ascites, encephalopathy, or variceal bleeding).
* Any other serious or active clinical condition or prior therapy that, in the opinion of the investigator, would make the individual unsuitable for the study or unable to comply with dosing requirements.
* Hepatitis C virus (HCV) antibody positive and detectable HCV RNA.
* Chronic hepatitis B virus (HBV) infection, as determined by either:

  * Positive HBV surface antigen and negative HBV surface antibody, regardless of HBV core antibody status, at the screening visit, or
  * Positive HBV core antibody and negative HBV surface antibody, regardless of HBV surface antigen status, at the screening visit.
* Hepatic transaminases (aspartate aminotransferase (AST) or alanine aminotransferase (ALT)) > 5 x upper limit of normal (ULN).
* Current alcohol or substance use judged by the investigator to potentially interfere with individual study compliance.
* Positive serum pregnancy test at screening or a positive pregnancy test prior to Day 1.
* Individuals with plan to breastfeed during the study period including the protocol-defined follow-up period.
* Requirement for ongoing therapy with or prior use of any prohibited medications listed in the protocol. Any prescription medications or over the counter medications, including herbal products, within 28 days prior to start of study drug dosing must be reviewed and approved by the sponsor, with the exception of vitamins and/or acetaminophen and/or ibuprofen.
* Any current or prior receipt of LA parenteral ARVs such as mAbs targeting HIV-1, injectable CAB, or injectable RPV, for treatment or prophylaxis (PrEP, PEP).

Substudy-01, Substudy-02, Substudy-03:

* Requirement for ongoing therapy with any prohibited medications listed in protocol.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2022-10-26 (Actual); Primary Completion 2024-02-17 (Actual); Study Completion 2024-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (42):
- United States (38):
  - Long Beach Education and Research Consultants,Substudy-03, Long Beach, California
  - Mills Clinical Research,Substudy-02, Los Angeles, California
  - Mills Clinical Research,Substudy-03, Los Angeles, California
  - Quest Clinical Research,Substudy-01, San Francisco, California
  - Quest Clinical Research,Substudy-02, San Francisco, California
  - Quest Clinical Research,Substudy-03, San Francisco, California
  - Yale University; School of Medicine; AIDS Program (Administrative & Study Supplies),Substudy-03, New Haven, Connecticut
  - Yale University,Substudy-02, New Haven, Connecticut
  - Washington Health Institute,Substudy-01, Washington D.C., District of Columbia
  - Washington Health Institute,Substudy-02, Washington D.C., District of Columbia
  - Washington Health Institute,Substudy-03, Washington D.C., District of Columbia
  - Midland Florida Clinical Research Center, LLC,Substudy-02, DeLand, Florida
  - Midland Florida Clinical Research, LLC,Substudy-03, DeLand, Florida
  - Midway Immunology and Research Center,Substudy-01, Ft. Pierce, Florida
  - Midway Immunology and Research Center,Substudy-02, Ft. Pierce, Florida
  - Midway Immunology and Research Center,Substudy-03, Ft. Pierce, Florida
  - Bliss Health,Substudy-02, Orlando, Florida
  - Bliss Health,Substudy-03, Orlando, Florida
  - Orlando Immunology Center,Substudy-01, Orlando, Florida
  - Orlando Immunology Center,Substudy-03, Orlando, Florida
  - Triple O Research Institute, P.A.,Substudy-01, West Palm Beach, Florida
  - Triple O Research Institute, P.A.,Substudy-03, West Palm Beach, Florida
  - Infectious Disease Specialists of Atlanta,Substudy-01, Decatur, Georgia
  - Indiana CTSI Clinical Research Center,Substudy-01, Indianapolis, Indiana
  - University of Cincinnati College of Medicine,Substudy-02, Cincinnati, Ohio
  - University of Cincinnati College of Medicine,Substudy-03, Cincinnati, Ohio
  - Central Texas Clinical Research,Substudy-01, Austin, Texas
  - Central Texas Clinical Research,Substudy-03, Austin, Texas
  - Prism Health North Texas,Substudy-02, Dallas, Texas
  - Prism Health North Texas,Substudy-03, Dallas, Texas
  - North Texas Infectious Diseases Consultant, P.A.,Substudy-02, Dallas, Texas
  - North Texas Infectious Diseases Consultants, P.A.,Substudy-03, Dallas, Texas
  - AXCES Research,Substudy-02, El Paso, Texas
  - AXES Research Group LLC,Substudy-03, El Paso, Texas
  - Therapeutic Concepts, PA,Substudy-02, Houston, Texas
  - Therapeutic Concepts, PA,Substudy-03, Houston, Texas
  - The Crofoot Research Center, Inc.,Substudy-01, Houston, Texas
  - MultiCare Rockwood Main Clinic- Research,Substudy-03, Spokane, Washington
- Instituto Dominicano de Estudio Virologicos - IDEV,Substudy-02, Santo Domingo, Dominican Republic
- Thailand (3):
  - The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT),Substudy-02, Bangkok
  - The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT),Substudy-03, Bangkok
  - Faculty of Medicine, Srinagarind Hospital, Khon Kaen University,Substudy-03, Khon Kaen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carl J. Fichtenbaum, Mezgebe Berhe, Jose Bordon, et al, Antiviral Activity, Safety, and Pharmacokinetics of GS-1720: A Novel Weekly Oral INSTI. Conference on Retroviruses and Opportunistic Infections, 2024, 3-6 March.
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-544-5905

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 100 participants were screened. Participants were enrolled at study sites in the United States, Thailand, and Dominican Republic.
Pre-assignment Details: Efficacy outcome measures (OM) included an additional cohort of Placebo. In this study, none of the participants received placebo. Placebo arm included 21 participants with HIV-1 from 3 other Gilead Phase 1b studies (GS-US-120-0104, GS-US-141-1219 (NCT02275065), and GS-US-200-4072 (NCT03739866)).
  Each bavtavirine, GS-1720, and GS-6212 cohort was compared to the pooled placebo cohort in the efficacy OMs #1, 2, and 17.
Groups:
- Substudy 01: Cohort 1: Bavtavirine 675 mg (High-Fat Meal): Participants received a single dose of bavtavirine 675 mg, tablets, orally, with a high-fat meal on Day 1. After assessments on Day 11 or upon early termination (ET), the participants initiated an oral regimen of bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF), or an alternative standard of care (SOC) antiretroviral therapy (ART) regimen (example integrase strand-transfer inhibitor (INSTI) + nucleoside reverse transcriptase inhibitor (NRTIs): Dolutegravir/abacavir/lamivudine (DTG/ABC/3TC) or DTG/3TC), orally up to Day 39.
- Substudy 01: Cohort 2: Bavtavirine 1200 mg (Low-Fat Meal): Participants received a single dose of bavtavirine 1200 mg, tablets, orally, with a low-fat meal on Day 1. After assessments on Day 11 or upon ET, the participants initiated an oral regimen of B/F/TAF, or an alternative SOC ART regimen (example INSTI + NRTIs: DTG/ABC/3TC or DTG/3TC), orally up to Day 39.
- Substudy 01: Cohort 3: Bavtavirine 900 mg (High-Fat Meal): Participants received a single dose of bavtavirine 900 mg, tablets, orally, with a high-fat meal on Days 1 and 2. After assessments on Day 11 or upon ET, the participants initiated an oral regimen of B/F/TAF, or an alternative SOC ART regimen (example INSTI + NRTIs: DTG/ABC/3TC or DTG/3TC), orally up to Day 39.
- Substudy 02: Cohort 1: GS-1720 450 mg: Participants received a single dose of GS-1720 450 mg, tablets, orally, on both Days 1 and 2 in fasted condition. After assessments on Day 11 or upon ET, the participants initiated an oral regimen of B/F/TAF, or an alternative SOC ART regimen (example INSTI + NRTIs: DTG/ABC/3TC or DTG/3TC), orally up to Day 60.
- Substudy 02: Cohort 2: GS-1720 150 mg: Participants received a single dose of GS-1720 150 mg, tablets, orally, on both Days 1 and 2 in fasted condition. After assessments on Day 11 or upon ET, the participants initiated an oral regimen of B/F/TAF, or an alternative SOC ART regimen (example INSTI + NRTIs: DTG/ABC/3TC or DTG/3TC), orally up to Day 60.
- Substudy 02: Cohort 3: GS-1720 30 mg: Participants received a single dose of GS-1720 30 mg, tablets, orally, on both Days 1 and 2 in fasted condition. After assessments on Day 11 or upon ET, the participants initiated an oral regimen of B/F/TAF, or an alternative SOC ART regimen (example INSTI + NRTIs: DTG/ABC/3TC or DTG/3TC), orally up to Day 60.
- Substudy 02: Cohort 4: GS-1720 900 mg: Participants received a single dose of GS-1720 900 mg, tablets, orally, on both Days 1 and 2 in fasted condition. After assessments on Day 11 or upon ET, the participants initiated an oral regimen of B/F/TAF, or an alternative SOC ART regimen (example INSTI + NRTIs: DTG/ABC/3TC or DTG/3TC), orally up to Day 60.
- Substudy 03: Cohort 1: GS- 6212 100 mg: Participants received GS-6212 100 mg tablet orally, twice daily on Days 1 through 10. After assessments on Day 11 or upon ET, the participants initiated an oral regimen of B/F/TAF, or an alternative SOC ART regimen (example INSTI + NRTIs: DTG/ABC/3TC or DTG/3TC), orally up to Day 25.
Period: Overall Study
Arm/Group | Substudy 01: Cohort 1: Bavtavirine 675 mg (High-Fat Meal) | Substudy 01: Cohort 2: Bavtavirine 1200 mg (Low-Fat Meal) | Substudy 01: Cohort 3: Bavtavirine 900 mg (High-Fat Meal) | Substudy 02: Cohort 1: GS-1720 450 mg | Substudy 02: Cohort 2: GS-1720 150 mg | Substudy 02: Cohort 3: GS-1720 30 mg | Substudy 02: Cohort 4: GS-1720 900 mg | Substudy 03: Cohort 1: GS- 6212 100 mg
Started | 6 | 6 | 1 | 7 | 7 | 7 | 7 | 8
Completed | 6 | 6 | 1 | 7 | 7 | 7 | 6 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who took at least 1 dose of the following: bavtavirine in Substudy 01; GS-1720 in Substudy 02 and GS-6212 in Substudy 03.
Groups:
- Substudy 01: Cohort 1: Bavtavirine 675 mg (High-Fat Meal): Participants received a single dose of bavtavirine 675 mg tablet, orally, with a high-fat meal on Day 1. After assessments on Day 11 or upon early termination (ET), the participants initiated an oral regimen of B/F/TAF, or an alternative SOC ART regimen (example INSTI + NRTIs: DTG/ABC/3TC or DTG/3TC), orally up to Day 39.
- Substudy 01: Cohort 2: Bavtavirine 1200 mg (Low-Fat Meal): Participants received a single dose of bavtavirine 1200 mg tablet, orally, with a low-fat meal on Day 1. After assessments on Day 11 or upon ET, the participants initiated an oral regimen of B/F/TAF, or an alternative SOC ART regimen (example INSTI + NRTIs: DTG/ABC/3TC or DTG/3TC), orally up to Day 39.
- Substudy 01: Cohort 3: Bavtavirine 900 mg (High-Fat Meal): Participants received a single dose of bavtavirine 900 mg tablet, orally, with a high-fat meal on Days 1 and 2. After assessments on Day 11 or upon ET, the participants initiated an oral regimen of B/F/TAF, or an alternative SOC ART regimen (example INSTI + NRTIs: DTG/ABC/3TC or DTG/3TC), orally up to Day 39.
- Substudy 02: Cohort 1: GS-1720 450 mg: Participants received a single dose of GS-1720 450 mg tablet, orally, on both Days 1 and 2 in fasted condition. After assessments on Day 11 or upon ET, the participants initiated an oral regimen of B/F/TAF, or an alternative SOC ART regimen (example INSTI + NRTIs: DTG/ABC/3TC or DTG/3TC), orally up to Day 60.
- Substudy 02: Cohort 2: GS-1720 150 mg: Participants received a single dose of GS-1720 150 mg tablet, orally, on both Days 1 and 2 in fasted condition. After assessments on Day 11 or upon ET, the participants initiated an oral regimen of B/F/TAF, or an alternative SOC ART regimen (example INSTI + NRTIs: DTG/ABC/3TC or DTG/3TC), orally up to Day 60.
- Substudy 02: Cohort 3: GS-1720 30 mg: Participants received a single dose of GS-1720 30 mg tablet, orally, on both Days 1 and 2 in fasted condition. After assessments on Day 11 or upon ET, the participants initiated an oral regimen of B/F/TAF, or an alternative SOC ART regimen (example INSTI + NRTIs: DTG/ABC/3TC or DTG/3TC), orally up to Day 60.
- Substudy 02: Cohort 4: GS-1720 900 mg: Participants received a single dose of GS-1720 900 mg tablet, orally, on both Days 1 and 2 in fasted condition. After assessments on Day 11 or upon ET, the participants initiated an oral regimen of B/F/TAF, or an alternative SOC ART regimen (example INSTI + NRTIs: DTG/ABC/3TC or DTG/3TC), orally up to Day 60.
- Substudy 03: Cohort 1: GS- 6212 100 mg: Participants received GS-6212 100 mg tablet, orally, twice daily on Days 1 through 10. After assessments on Day 11 or upon ET, the participants initiated an oral regimen of B/F/TAF, or an alternative SOC ART regimen (example INSTI + NRTIs: DTG/ABC/3TC or DTG/3TC), orally up to Day 25.
- Total: Total of all reporting groups
Arm/Group | Substudy 01: Cohort 1: Bavtavirine 675 mg (High-Fat Meal) | Substudy 01: Cohort 2: Bavtavirine 1200 mg (Low-Fat Meal) | Substudy 01: Cohort 3: Bavtavirine 900 mg (High-Fat Meal) | Substudy 02: Cohort 1: GS-1720 450 mg | Substudy 02: Cohort 2: GS-1720 150 mg | Substudy 02: Cohort 3: GS-1720 30 mg | Substudy 02: Cohort 4: GS-1720 900 mg | Substudy 03: Cohort 1: GS- 6212 100 mg | Total
Number analyzed (Participants) | 6 | 6 | 1 | 7 | 7 | 7 | 7 | 8 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
  Between 18 and 65 years | 5 | 6 | 1 | 7 | 7 | 6 | 7 | 8 | 47
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (9.5) | 38 (13.9) | 31 (NA) — Standard deviation could not be calculated for one participant. | 35 (13.9) | 42 (13.5) | 39 (13.0) | 32 (6.5) | 33 (11.9) | 36 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 8
  Male | 4 | 5 | 0 | 6 | 6 | 6 | 7 | 7 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 0 | 2 | 2 | 4 | 5 | 2 | 19
  Not Hispanic or Latino | 4 | 4 | 1 | 5 | 5 | 3 | 2 | 6 | 30
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2
  Black or African American | 3 | 3 | 1 | 0 | 3 | 3 | 0 | 3 | 16
  White | 2 | 3 | 0 | 3 | 3 | 1 | 2 | 4 | 18
  More than one race | 1 | 0 | 0 | 2 | 0 | 2 | 3 | 0 | 8
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 6 | 1 | 7 | 7 | 5 | 3 | 7 | 42
  Dominican Republic | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 5
  Thailand | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Substudies 01, 02 and 03: Change From Baseline in Plasma Human Immunodeficiency Virus (HIV)-1 Ribonucleic Acid (RNA) (log10 Copies/mL) at Day 11 Relative to Historical Placebo Data
Time Frame: Baseline, Day 11
Population: Participants in the Full Analysis Set with data available were analyzed. The Full Analysis Set included all participants who were enrolled and received full dose(s) of study drugs bavtavirine, GS-1720 and GS-6212 in these substudies.
  The placebo arm included pooled data from participants who received placebo in 3 historical Gilead HIV-1 phase 1b studies (GS-US-120-0104, GS-US-141-1219, and GS-US-200-4072) for HIV-1 efficacy parameters only.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Groups:
- Substudy 01: Cohort 1: Bavtavirine 675 mg (High-Fat Meal): Participants received a single dose of bavtavirine 675 mg, tablets, orally, with a high-fat meal on Day 1. After assessments on Day 11 or upon early termination (ET), the participants initiated an oral regimen of B/F/TAF, or an alternative SOC ART regimen (example INSTI + NRTIs: DTG/ABC/3TC or DTG/3TC), orally up to Day 39.
- Substudy 03: Cohort 1: GS- 6212 100 mg: Participants received GS-6212 100 mg tablet orally twice daily on Days 1 through 10. After assessments on Day 11 or upon ET, the participants initiated an oral regimen of B/F/TAF, or an alternative SOC ART regimen (example INSTI + NRTIs: DTG/ABC/3TC or DTG/3TC), orally up to Day 25.
- Placebo: Historical data for the placebo participants from 3 sponsor Phase 1b studies (GS-US-120-0104, GS-US-141-1219, and GS-US-200-4072) were combined to form a single placebo group for the purpose of analysis. For Study GS-US-200-4072, HIV-1 RNA (log10 copies/mL) collected on Day 10 was used for "Day 11", since HIV-1 RNA was not collected on Day 11 for this study. Each GS-1720 cohort was compared to the pooled placebo group with respect to the change from baseline in plasma HIV-1 RNA (log10 copies/mL) on Day 11.
Arm/Group | Substudy 01: Cohort 1: Bavtavirine 675 mg (High-Fat Meal) | Substudy 01: Cohort 2: Bavtavirine 1200 mg (Low-Fat Meal) | Substudy 01: Cohort 3: Bavtavirine 900 mg (High-Fat Meal) | Substudy 02: Cohort 1: GS-1720 450 mg | Substudy 02: Cohort 2: GS-1720 150 mg | Substudy 02: Cohort 3: GS-1720 30 mg | Substudy 02: Cohort 4: GS-1720 900 mg | Substudy 03: Cohort 1: GS- 6212 100 mg | Placebo
Number analyzed (Participants) | 6 | 6 | 1 | 7 | 7 | 7 | 7 | 8 | 21
log10 copies/mL
  Baseline | 4.68 (0.517) | 4.68 (0.488) | 4.27 (NA) — Standard deviation could not be calculated for one participant. | 5.16 (0.562) | 4.72 (0.362) | 4.52 (0.565) | 4.93 (0.366) | 4.41 (0.850) | 4.43 (0.508)
  Change from Baseline at Day 11: number analyzed (Participants) | 6 | 5 | 1 | 7 | 7 | 7 | 7 | 6 | 21
  Change from Baseline at Day 11 | -1.40 (0.454) | -1.46 (0.690) | -1.54 (NA) — Standard deviation could not be calculated for one participant. | -2.44 (0.425) | -2.18 (0.199) | -1.74 (0.766) | -2.37 (0.509) | -2.43 (0.698) | 0.01 (0.338)
Statistical Analysis 1: Comparison: Substudy 01: Cohort 1: Bavtavirine 675 mg (High-Fat Meal) vs Placebo; Test type: Superiority; p < 0.0001, t-test, 2 sided — P-value was calculated from two-sided t-test
Statistical Analysis 2: Comparison: Substudy 01: Cohort 2: Bavtavirine 1200 mg (Low-Fat Meal) vs Placebo; Test type: Superiority; p < 0.0001, t-test, 2 sided — P-value was calculated from two-sided t-test
Statistical Analysis 3: Comparison: Substudy 01: Cohort 3: Bavtavirine 900 mg (High-Fat Meal) vs Placebo; Test type: Superiority; p = 0.0013, t-test, 2 sided — P-value was calculated from two-sided t-test
Statistical Analysis 4: Comparison: Substudy 02: Cohort 1: GS-1720 450 mg vs Placebo; Test type: Superiority; p < 0.0001, t-test, 2 sided — P-value was calculated from two-sided t-test
Statistical Analysis 5: Comparison: Substudy 02: Cohort 2: GS-1720 150 mg vs Placebo; Test type: Superiority; p < 0.0001, t-test, 2 sided — P-value was calculated from two-sided t-test
Statistical Analysis 6: Comparison: Substudy 02: Cohort 3: GS-1720 30 mg vs Placebo; Test type: Superiority; p < 0.0001, t-test, 2 sided — P-value was calculated from two-sided t-test
Statistical Analysis 7: Comparison: Substudy 02: Cohort 4: GS-1720 900 mg vs Placebo; Test type: Superiority; p < 0.0001, t-test, 2 sided — P-value was calculated from two-sided t-test
Statistical Analysis 8: Comparison: Substudy 03: Cohort 1: GS- 6212 100 mg vs Placebo; Test type: Superiority; p < 0.0001, t-test, 2 sided — P-value was calculated from two-sided t-test

2. Secondary Outcome: Substudies 01, 02 and 03: Change From Baseline in Plasma HIV-1 RNA (log10 Copies/mL) at Day 8 Relative to Historical Placebo Data
Time Frame: Baseline, Day 8
Population: Participants in the Full Analysis Set with available data were analyzed. The placebo arm included pooled data from participants who received placebo in 3 historical Gilead HIV-1 phase 1b studies (GS-US-120-0104, GS-US-141-1219, and GS-US-200-4072) for HIV-1 efficacy parameters only.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Substudy 01: Cohort 1: Bavtavirine 675 mg (High-Fat Meal) | Substudy 01: Cohort 2: Bavtavirine 1200 mg (Low-Fat Meal) | Substudy 01: Cohort 3: Bavtavirine 900 mg (High-Fat Meal) | Substudy 02: Cohort 1: GS-1720 450 mg | Substudy 02: Cohort 2: GS-1720 150 mg | Substudy 02: Cohort 3: GS-1720 30 mg | Substudy 02: Cohort 4: GS-1720 900 mg | Substudy 03: Cohort 1: GS- 6212 100 mg | Placebo
Number analyzed (Participants) | 6 | 6 | 1 | 7 | 7 | 7 | 7 | 8 | 21
log10 copies/mL
  Baseline | 4.68 (0.517) | 4.68 (0.488) | 4.27 (NA) — Standard deviation could not be calculated for one participant. | 5.16 (0.562) | 4.72 (0.362) | 4.52 (0.565) | 4.93 (0.366) | 4.41 (0.850) | 4.43 (0.508)
  Change from Baseline at Day 8: number analyzed (Participants) | 6 | 5 | 1 | 7 | 7 | 7 | 7 | 6 | 20
  Change from Baseline at Day 8 | -1.49 (0.239) | -1.54 (0.497) | -1.51 (NA) — Standard deviation could not be calculated for one participant. | -2.04 (0.346) | -1.76 (0.185) | -1.67 (0.326) | -1.98 (0.249) | -2.10 (0.417) | 0.01 (0.297)
Statistical Analysis 1: Comparison: Substudy 01: Cohort 1: Bavtavirine 675 mg (High-Fat Meal) vs Placebo; Test type: Superiority; p < 0.0001, t-test, 2 sided — P-value was calculated from two-sided t-test
Statistical Analysis 2: Comparison: Substudy 01: Cohort 2: Bavtavirine 1200 mg (Low-Fat Meal) vs Placebo; Test type: Superiority; p < 0.0001, t-test, 2 sided — P-value was calculated from two-sided t-test
Statistical Analysis 3: Comparison: Substudy 01: Cohort 3: Bavtavirine 900 mg (High-Fat Meal) vs Placebo; Test type: Superiority; p < 0.0001, t-test, 2 sided — P-value was calculated from two-sided t-test
Statistical Analysis 4: Comparison: Substudy 02: Cohort 1: GS-1720 450 mg vs Placebo; Test type: Superiority; p < 0.0001, t-test, 2 sided — P-value was calculated from two-sided t-test
Statistical Analysis 5: Comparison: Substudy 02: Cohort 2: GS-1720 150 mg vs Placebo; Test type: Superiority; p < 0.0001, t-test, 2 sided — P-value was calculated from two-sided t-test
Statistical Analysis 6: Comparison: Substudy 02: Cohort 3: GS-1720 30 mg vs Placebo; Test type: Superiority; p < 0.0001, t-test, 2 sided — P-value was calculated from two-sided t-test
Statistical Analysis 7: Comparison: Substudy 02: Cohort 4: GS-1720 900 mg vs Placebo; Test type: Superiority; p < 0.0001, t-test, 2 sided — P-value was calculated from two-sided t-test
Statistical Analysis 8: Comparison: Substudy 03: Cohort 1: GS- 6212 100 mg vs Placebo; Test type: Superiority; p < 0.0001, t-test, 2 sided — P-value was calculated from two-sided t-test

3. Secondary Outcome: Substudies 01, 02 and 03: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. TEAEs were defined as any AEs with an onset date on or after the study drug start date.
  Percentages were rounded-off.
Time Frame: First dose up to last dose (Substudy 01: Up to Day 39; Substudy 02: Up to Day 60; Substudy 03: Up to Day 25)
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Groups:
- Substudy 03: Cohort 1: GS- 6212 100 mg: Participants received GS-6212 100 mg tablets orally twice daily on Days 1 through 10. After assessments on Day 11 or upon ET, the participants initiated an oral regimen of B/F/TAF, or an alternative SOC ART regimen (example INSTI + NRTIs: DTG/ABC/3TC or DTG/3TC), orally up to Day 25.
Arm/Group | Substudy 01: Cohort 1: Bavtavirine 675 mg (High-Fat Meal) | Substudy 01: Cohort 2: Bavtavirine 1200 mg (Low-Fat Meal) | Substudy 01: Cohort 3: Bavtavirine 900 mg (High-Fat Meal) | Substudy 02: Cohort 1: GS-1720 450 mg | Substudy 02: Cohort 2: GS-1720 150 mg | Substudy 02: Cohort 3: GS-1720 30 mg | Substudy 02: Cohort 4: GS-1720 900 mg | Substudy 03: Cohort 1: GS- 6212 100 mg
Number analyzed (Participants) | 6 | 6 | 1 | 7 | 7 | 7 | 7 | 8
percentage of participants | 50.0 | 16.7 | 100 | 42.9 | 85.7 | 85.7 | 71.4 | 75.0

4. Secondary Outcome: Substudies 01, 02 and 03: Percentage of Participants With Graded Laboratory Abnormalities
Description: Treatment-emergent laboratory abnormalities were defined as values that increased at least 1 toxicity grade from baseline at any time postbaseline. Laboratory abnormalities were graded using Division of AIDS (DAIDS) scale with grade 0 to 4 where 0 = no grade; 1 = mild, 2 = moderate, 3 = severe; 4 = potentially life-threatening. Participants with at least a 1 grade increased from baseline for an individual laboratory test where the maximum post baseline laboratory abnormality was 1) grade 1 or higher and 2) grade 3 or higher were reported. The maximum postbaseline toxicity grade across all tests for an individual participant was used in analysis. Percentages were rounded-off.
Time Frame: First dose up to last dose (Substudy 01: Up to Day 39; Substudy 02: Up to Day 60; Substudy 03: Up to Day 25)
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Groups:
- Substudy 03: Cohort 1: GS- 6212 100 mg: Participants received GS-6212 100 mg, tablet, orally, twice daily on Days 1 through 10. After assessments on Day 11 or upon ET, the participants initiated an oral regimen of B/F/TAF, or an alternative SOC ART regimen (example INSTI + NRTIs: DTG/ABC/3TC or DTG/3TC), orally up to Day 25.
Arm/Group | Substudy 01: Cohort 1: Bavtavirine 675 mg (High-Fat Meal) | Substudy 01: Cohort 2: Bavtavirine 1200 mg (Low-Fat Meal) | Substudy 01: Cohort 3: Bavtavirine 900 mg (High-Fat Meal) | Substudy 02: Cohort 1: GS-1720 450 mg | Substudy 02: Cohort 2: GS-1720 150 mg | Substudy 02: Cohort 3: GS-1720 30 mg | Substudy 02: Cohort 4: GS-1720 900 mg | Substudy 03: Cohort 1: GS- 6212 100 mg
Number analyzed (Participants) | 6 | 6 | 1 | 7 | 7 | 7 | 7 | 8
percentage of participants
  Grade 1 or Higher | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 87.5
  Grade 3 or Higher | 16.7 | 66.7 | 0 | 0 | 14.3 | 14.3 | 0 | 0

5. Secondary Outcome: Substudy 01: Pharmacokinetic (PK) Parameter: Cmax of Bavtavirine
Description: Cmax was defined as the maximum observed concentration of drug.
Time Frame: Cohorts 1, 2 and 3 (Day 1: Predose, 0.5, 1, 2, 3, 4, 5, 6, 8, and 12 hours postdose); Cohort 3: Day 2: Predose, 0.5, 1, 2, 3, 4, 5, 6, and 8 hours postdose
Population: Participants in PK Analysis Set in Substudy 01 were analyzed. The PK Analysis Set included all participants who were enrolled in the study, received at least 1 dose of study drug, and had at least 1 non-missing post baseline concentration value for bavtavirine. Per pre-specified analysis, Cmax at Day 2 was calculated only for Cohort 3.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Substudy 01: Cohort 1: Bavtavirine 675 mg (High-Fat Meal) | Substudy 01: Cohort 2: Bavtavirine 1200 mg (Low-Fat Meal) | Substudy 01: Cohort 3: Bavtavirine 900 mg (High-Fat Meal)
Number analyzed (Participants) | 6 | 6 | 1
ng/mL
  Cmax (Day 1) | 685 (172) | 700 (364) | 565 (NA) — Standard deviation could not be calculated for one participant.
  Cmax (Day 2): number analyzed (Participants) | 0 | 0 | 1
  Cmax (Day 2) |  |  | 1160 (NA) — Standard deviation could not be calculated for one participant.

6. Secondary Outcome: Substudy 01: PK Parameter: AUC of Bavtavirine
Description: AUC was defined as the area under the concentration versus time curve.
Time Frame: Day 1 up to Day 11
Population: Participants in the PK Analysis Set in Substudy 01 were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Substudy 01: Cohort 1: Bavtavirine 675 mg (High-Fat Meal) | Substudy 01: Cohort 2: Bavtavirine 1200 mg (Low-Fat Meal) | Substudy 01: Cohort 3: Bavtavirine 900 mg (High-Fat Meal)
Number analyzed (Participants) | 6 | 6 | 1
h*ng/mL
  AUC (Days 1-8) | 33,300 (10300) | 24,300 (13700) | 71,400 (NA) — Standard deviation could not be calculated for one participant.
  AUC (Days 1-11) | 38,800 (11800) | 28,300 (16100) | 89,100 (NA) — Standard deviation could not be calculated for one participant.

7. Secondary Outcome: Substudy 01: PK Parameter: Plasma Concentration of Bavtavirine
Time Frame: Days 8 and 11
Population: Participants in the PK Analysis Set in Substudy 01 with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Substudy 01: Cohort 1: Bavtavirine 675 mg (High-Fat Meal) | Substudy 01: Cohort 2: Bavtavirine 1200 mg (Low-Fat Meal) | Substudy 01: Cohort 3: Bavtavirine 900 mg (High-Fat Meal)
Number analyzed (Participants) | 6 | 6 | 1
ng/mL
  Day 8: number analyzed (Participants) | 6 | 5 | 1
  Day 8 | 94.5 (36.8) | 64.8 (44.7) | 250 (NA) — Standard deviation could not be calculated for one participant.
  Day 11 | 61.2 (26.0) | 44.6 (32.8) | 202 (NA) — Standard deviation could not be calculated for one participant.

8. Secondary Outcome: Substudy 02: PK Parameter: Cmax of GS-1720
Description: Cmax was defined as the maximum observed concentration of drug.
Time Frame: Days 1 and 2: Predose, 0.5, 1, 2, 3, 4, 5, 6, 8 and (optional) 12 hours postdose
Population: Participants in the PK Analysis Set in Substudy 02 with available data were analyzed.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Substudy 02: Cohort 1: GS-1720 450 mg | Substudy 02: Cohort 2: GS-1720 150 mg | Substudy 02: Cohort 3: GS-1720 30 mg | Substudy 02: Cohort 4: GS-1720 900 mg
Number analyzed (Participants) | 7 | 7 | 7 | 7
µg/mL
  Cmax (Day 1) | 17.2 (8.37) | 9.77 (3.09) | 3.00 (0.691) | 33.7 (11.6)
  Cmax (Day 2): number analyzed (Participants) | 7 | 7 | 6 | 7
  Cmax (Day 2) | 30.8 (10.7) | 15.6 (5.59) | 5.39 (1.48) | 48.3 (9.85)

9. Secondary Outcome: Substudy 02: PK Parameter: AUC of GS-1720
Description: AUC was defined as the area under the concentration versus time curve.
Time Frame: Day 1 up to Day 11
Population: Participants in the PK Analysis Set in Substudy 02 were analyzed.
Measure: Mean (Standard Deviation); unit: h*µg/mL
Arm/Group | Substudy 02: Cohort 1: GS-1720 450 mg | Substudy 02: Cohort 2: GS-1720 150 mg | Substudy 02: Cohort 3: GS-1720 30 mg | Substudy 02: Cohort 4: GS-1720 900 mg
Number analyzed (Participants) | 7 | 7 | 7 | 7
h*µg/mL
  AUC (Day 8) | 2790 (1060) | 1670 (780) | 503 (134) | 4960 (1360)
  AUC (Day 11) | 3540 (1330) | 2160 (1020) | 648 (169) | 6430 (1740)

10. Secondary Outcome: Substudy 02: PK Parameter: Plasma Concentration of GS-1720
Time Frame: Days 8 and 11
Population: Participants in the PK Analysis Set in Substudy 02 were analyzed.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Substudy 02: Cohort 1: GS-1720 450 mg | Substudy 02: Cohort 2: GS-1720 150 mg | Substudy 02: Cohort 3: GS-1720 30 mg | Substudy 02: Cohort 4: GS-1720 900 mg
Number analyzed (Participants) | 7 | 7 | 7 | 7
µg/mL
  Day 8 | 12.2 (4.21) | 7.44 (3.65) | 2.59 (0.868) | 22.7 (4.94)
  Day 11 | 8.78 (4.15) | 5.87 (2.98) | 1.64 (0.376) | 18.4 (4.75)

11. Secondary Outcome: Substudy 03: PK Parameter: Cmax of GS-6212
Description: Cmax was defined as the maximum observed concentration of drug.
Time Frame: Days 1 and 10 (Predose, 0.25, 0.5, 1, 2, 3, 4, 6, 8 and (optional) 12 hours postdose)
Population: Participants in the PK Analysis Set in Substudy 03 with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Substudy 03: Cohort 1: GS- 6212 100 mg
Number analyzed (Participants) | 8
ng/mL
  Cmax (Day 1) | 1590 (641)
  Cmax (Day 10): number analyzed (Participants) | 6
  Cmax (Day 10) | 1550 (621)

12. Secondary Outcome: Substudy 03: PK Parameter: AUC0-8h of GS-6212
Description: AUC0-8h was defined as the area under the concentration versus time curve spanning from 0 to 8 hours post dose.
Time Frame: Days 1 and 10 (Predose, 0.25, 0.5, 1, 2, 3, 4, 6, 8 and (optional) 12 hours postdose)
Population: Participants in the PK Analysis Set in Substudy 03 with available data were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- Substudy 03: Cohort 1: GS- 6212 100 mg: Participants received GS-6212 100 mg, tablet, orally, twice daily on Days 1 through 10. After assessments on Day 11 or upon ET, the participants initiated an oral regimen of B/F/TAF, or an alternative SOC ART regimen (orally DTG/ABC/3TC or DTG/3TC), orally up to Day 25.
Arm/Group | Substudy 03: Cohort 1: GS- 6212 100 mg
Number analyzed (Participants) | 8
h*ng/mL
  AUC0-8h (Day 1) | 5030 (2190)
  AUC0-8h (Day 10): number analyzed (Participants) | 6
  AUC0-8h (Day 10) | 5700 (2300)

13. Secondary Outcome: Substudy 03: PK Parameter: AUCtau of GS-6212
Description: AUCtau was defined as the area under the curve from time zero to end of dosing interval.
Time Frame: Day 10 (Parameter estimated based on observed data from 0 to 8 hours postdose)
Population: Participants in the PK Analysis Set in Substudy 03 with available data were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Substudy 03: Cohort 1: GS- 6212 100 mg
Number analyzed (Participants) | 6
h*ng/mL | 6450 (2370)

14. Secondary Outcome: Substudy 03: PK Parameter: Plasma Concentration of GS-6212
Time Frame: Days 1 and 10: 8 hours postdose
Population: Participants in the PK Analysis Set in Substudy 03 with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Substudy 03: Cohort 1: GS- 6212 100 mg
Number analyzed (Participants) | 8
ng/mL
  C8h (Day 1) | 221 (165)
  C8h (Day 10): number analyzed (Participants) | 6
  C8h (Day 10) | 260 (194)

15. Secondary Outcome: Substudy 03: PK Parameter: Ctrough of GS-6212 (Day 10)
Description: Ctrough was defined as concentration at the end of the dosing interval.
Time Frame: Day 10 (Parameter estimated based on observed data from 0 to 8 hours postdose)
Population: Participants in the PK Analysis Set in Substudy 03 with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Substudy 03: Cohort 1: GS- 6212 100 mg
Number analyzed (Participants) | 6
ng/mL | 140 (207)

16. Secondary Outcome: Substudy 03: PK Parameter: Cavg of GS-6212 (Day 10)
Description: Cavg was defined as average plasma concentration during dose administration.
Time Frame: Day 10 (predose to 8 hours postdose)
Population: Participants in the PK Analysis Set in Substudy 03 with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Substudy 03: Cohort 1: GS- 6212 100 mg
Number analyzed (Participants) | 6
ng/mL | 538 (198)

17. Secondary Outcome: Substudies 01, 02 and 03: Percentage of Participants at Any Measurement Achieving HIV-1 RNA < 50 Copies/mL by Day 11 at Each Dose Level
Description: Percentages were rounded-off.
Time Frame: Up to Day 11
Population: Participants in the Full Analysis Set were analyzed. The placebo arm included pooled data from participants who received placebo in 3 historical Gilead HIV-1 phase 1b studies (GS-US-120-0104, GS-US-141-1219, and GS-US-200-4072) for HIV-1 efficacy parameters only.
Measure: Number; unit: percentage of participants
Groups:
- Substudy 03: Cohort 1: GS- 6212 100 mg BID: Participants received GS-6212 100 mg, tablet, orally, twice daily on Days 1 through 10. After assessments on Day 11 or upon ET, the participants initiated an oral regimen of B/F/TAF, or an alternative SOC ART regimen (example INSTI + NRTIs: DTG/ABC/3TC or DTG/3TC), orally up to Day 25.
Arm/Group | Substudy 01: Cohort 1: Bavtavirine 675 mg (High-Fat Meal) | Substudy 01: Cohort 2: Bavtavirine 1200 mg (Low-Fat Meal) | Substudy 01: Cohort 3: Bavtavirine 900 mg (High-Fat Meal) | Substudy 02: Cohort 1: GS-1720 450 mg | Substudy 02: Cohort 2: GS-1720 150 mg | Substudy 02: Cohort 3: GS-1720 30 mg | Substudy 02: Cohort 4: GS-1720 900 mg | Substudy 03: Cohort 1: GS- 6212 100 mg BID | Placebo
Number analyzed (Participants) | 6 | 6 | 1 | 7 | 7 | 7 | 7 | 8 | 21
percentage of participants | 0 | 0 | 0 | 0 | 0 | 28.6 | 0 | 37.5 | 0

18. Secondary Outcome: Substudies 01, 02 and 03: Percentage of Participants With Emergence of Viral Resistance to the ARV Class of the Given Drug
Description: The antiretroviral (ARV) class of given drugs would be BVY or NNRTIs (Substudy 01) or INSTIs (Substudy 02) or INSTIs (Substudy 03).
  Percentages were rounded-off.
Time Frame: Up to Day 11
Population: Participant in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Substudy 01: Cohort 1: Bavtavirine 675 mg (High-Fat Meal) | Substudy 01: Cohort 2: Bavtavirine 1200 mg (Low-Fat Meal) | Substudy 01: Cohort 3: Bavtavirine 900 mg (High-Fat Meal) | Substudy 02: Cohort 1: GS-1720 450 mg | Substudy 02: Cohort 2: GS-1720 150 mg | Substudy 02: Cohort 3: GS-1720 30 mg | Substudy 02: Cohort 4: GS-1720 900 mg | Substudy 03: Cohort 1: GS- 6212 100 mg BID
Number analyzed (Participants) | 6 | 6 | 1 | 7 | 7 | 7 | 7 | 8
percentage of participants | 33.0 | 16.6 | 0 | 0 | 0 | 0 | 0 | 0

19. Secondary Outcome: Substudy 01: Maximum Inhibitory Quotient (IQ) of Bavtavirine by Mean Plasma Concentration (Ct) up to Day 11
Description: Inhibitory quotient was calculated as the ratio of bavtavirine in vivo exposure to in vitro plasma concentration. IQ is defined as paEC95. paEC95 = protein-adjusted effective concentration to achieve 95% effective inhibition. The IQ ≥ 2 indicated higher reduction in viral load with less rebound.
Time Frame: Up to Day 11
Population: The PK/PD Analysis Set included all participants who were in the Full Analysis Set and have both nonmissing Ct (and/or AUC) of study drug and the change from baseline at Day 11 in plasma HIV-1 RNA (log10 copies/mL).
Measure: Number; unit: ratio
Arm/Group | Substudy 01: Cohort 1: Bavtavirine 675 mg (High-Fat Meal) | Substudy 01: Cohort 2: Bavtavirine 1200 mg (Low-Fat Meal) | Substudy 01: Cohort 3: Bavtavirine 900 mg (High-Fat Meal)
Number analyzed (Participants) | 6 | 6 | 1
ratio | 5 | 5 | 5

20. Secondary Outcome: Substudy 02: Inhibitory Quotient (IQ) of GS-1720 by Mean Plasma Concentration (Ct) at Day 11
Description: Inhibitory quotient was calculated as the ratio of GS-1720 in vivo exposure to in vitro plasma concentration. IQ is defined as paEC95. paEC95 = protein-adjusted effective concentration to achieve 95% effective inhibition. The IQ ≥ 2 indicated higher reduction in viral load with less rebound.
Time Frame: Day 11
Population: Participants in the PK/PD Analysis Set were analyzed.
Measure: Number; unit: ratio
Arm/Group | Substudy 02: Cohort 1: GS-1720 450 mg | Substudy 02: Cohort 2: GS-1720 150 mg | Substudy 02: Cohort 3: GS-1720 30 mg | Substudy 02: Cohort 4: GS-1720 900 mg
Number analyzed (Participants) | 7 | 7 | 7 | 7
ratio | 4.5 | 3 | 0.8 | 9.5

21. Secondary Outcome: Substudy 03: Inhibitory Quotient (IQ) of GS-6212 by Ctrough at Day 11
Description: Ctrough is the plasma concentration of the drug just before the next dose. Inhibitory quotient was calculated as the ratio of GS-1720 in vivo exposure to in vitro Ctrough. IQ is defined as paEC95. paEC95 = protein-adjusted effective concentration to achieve 95% effective inhibition. The IQ ≥ 2 indicated higher reduction in viral load with less rebound.
Time Frame: Day 11
Population: Participants in the PK/PD Analysis Set with available data were analyzed.
Measure: Number; unit: ratio
Arm/Group | Substudy 03: Cohort 1: GS- 6212 100 mg
Number analyzed (Participants) | 3
ratio | 6.5

ADVERSE EVENTS:
Time Frame: Substudy 01: Up to Day 39; Substudy 02: Up to Up to Day 60; Substudy 03: Up to Day 25
Description: All-Cause Mortality: All Enrolled Analysis Set included all participants who received a study participant ID number in the study after screening.
  Adverse Events: The Safety Analysis Set included all participants who took at least 1 dose of bavtavirine, GS-1720, and GS-6212 in this study.
Arm/Group | Substudy 01: Cohort 1: Bavtavirine 675 mg (High-Fat Meal) | Substudy 01: Cohort 2: Bavtavirine 1200 mg (Low-Fat Meal) | Substudy 01: Cohort 3: Bavtavirine 900 mg (High-Fat Meal) | Substudy 02: Cohort 1: GS-1720 450 mg | Substudy 02: Cohort 2: GS-1720 150 mg | Substudy 02: Cohort 3: GS-1720 30 mg | Substudy 02: Cohort 4: GS-1720 900 mg | Substudy 03: Cohort 1: GS- 6212 100 mg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/1 | 0/7 | 0/7 | 0/7 | 0/7 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/6 | 0/1 | 0/7 | 1/7 | 0/7 | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 3/6 | 0/6 | 1/1 | 3/7 | 6/7 | 6/7 | 5/7 | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Substudy 01: Cohort 1: Bavtavirine 675 mg (High-Fat Meal) (N=6) | Substudy 01: Cohort 2: Bavtavirine 1200 mg (Low-Fat Meal) (N=6) | Substudy 01: Cohort 3: Bavtavirine 900 mg (High-Fat Meal) (N=1) | Substudy 02: Cohort 1: GS-1720 450 mg (N=7) | Substudy 02: Cohort 2: GS-1720 150 mg (N=7) | Substudy 02: Cohort 3: GS-1720 30 mg (N=7) | Substudy 02: Cohort 4: GS-1720 900 mg (N=7) | Substudy 03: Cohort 1: GS- 6212 100 mg (N=8)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Suicidal behaviour (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Substudy 01: Cohort 1: Bavtavirine 675 mg (High-Fat Meal) (N=6) | Substudy 01: Cohort 2: Bavtavirine 1200 mg (Low-Fat Meal) (N=6) | Substudy 01: Cohort 3: Bavtavirine 900 mg (High-Fat Meal) (N=1) | Substudy 02: Cohort 1: GS-1720 450 mg (N=7) | Substudy 02: Cohort 2: GS-1720 150 mg (N=7) | Substudy 02: Cohort 3: GS-1720 30 mg (N=7) | Substudy 02: Cohort 4: GS-1720 900 mg (N=7) | Substudy 03: Cohort 1: GS- 6212 100 mg (N=8)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hangover (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anal fistula infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Body tinea (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Conjunctivitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pyuria (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Syphilis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Procedural headache (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Creatinine renal clearance abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Electrocardiogram ST segment abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Electrocardiogram T wave abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neisseria test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sars-cov-2 test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Device loosening (Product Issues) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Terminal insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years.

DOCUMENTS (6):
  • Study Protocol: Substudy 01 Protocol Amendment 01 (2022-09-27): https://cdn.clinicaltrials.gov/large-docs/07/NCT05585307/Prot_000.pdf
  • Study Protocol: Substudy 02 Protocol Amendment 02 (2023-05-05): https://cdn.clinicaltrials.gov/large-docs/07/NCT05585307/Prot_001.pdf
  • Study Protocol: Substudy 03 Protocol Amendment 01 (2023-08-18): https://cdn.clinicaltrials.gov/large-docs/07/NCT05585307/Prot_002.pdf
  • Statistical Analysis Plan: Substudy 01 Statistical Analysis Plan (2023-09-15): https://cdn.clinicaltrials.gov/large-docs/07/NCT05585307/SAP_003.pdf
  • Statistical Analysis Plan: Substudy 02 Statistical Analysis Plan (2024-05-16): https://cdn.clinicaltrials.gov/large-docs/07/NCT05585307/SAP_004.pdf
  • Statistical Analysis Plan: Substudy 03 Statistical Analysis Plan (2024-08-27): https://cdn.clinicaltrials.gov/large-docs/07/NCT05585307/SAP_005.pdf